CLINICAL TRIAL: NCT06812676
Title: Virtual Reality Induced Analgesia for Nasal Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Virtual Reality
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-12

CONDITIONS: Sinus Disease; Rhinitis; Turbinate; Hypertrophy Mucous Membrane; Deviated Nasal Septum Acquired; Deviated Nasal Septum - Congenital
Keywords: Virtual Reality; Nasal Procedures; Nasal Endoscopy; Otolaryngology; Pain Management; Non-pharmacological Intervention; Quality of Care
MeSH Terms: conditions — Paranasal Sinus Diseases; Rhinitis; Agnosia

STUDY DESIGN:
Intervention Model Description: Enrolled patients will be given a VR headset to wear during the nasal endoscopic procedure at the clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Arm (Experimental): The VR group will wear the VR
  Interventions: Device: Virtual Reality Goggles
- Standard of care Arm (No Intervention): patients will receive the standard of care

INTERVENTIONS:
Device: Virtual Reality Goggles — The VR group will be given a VR headset to wear during the nasal endoscopic procedure at the clinic.
  Arms: VR Arm

SUMMARY:
In-office nasal procedures can cause pain and discomfort to otolaryngology patients. While local anesthesia is the mainstay choice for main management, patients may have allergies or contraindications to the anesthetic agents used. Moreover, some procedures may not require it, or patients may benefit from additional pain management techniques. The immersive experience of Virtual Reality (VR) could benefit those patients by utilizing visual stimuli to reduce pain perception in the body. This study aims to investigate the efficacy of VR for pain management, and to assess the overall satisfaction of patients. If proven effective, VR could provide a safe non-pharmacological treatment for reducing pain and improving comfort of patients, thus raising the quality of care in otolaryngology clinic.

DETAILED DESCRIPTION:
Otolaryngology patients undergo routine office-based procedures such as nasal endoscopy, which may trigger distress, pain, and anxiety (1). This anxiety can, in turn, further exacerbate patients' perception of pain, which may require medication to alleviate. Minimizing unnecessary pharmacotherapy and reducing the risks associated with the side effects of pharmacologic treatments are of utmost importance. In addition, due to the ongoing opioid crisis, there is an urgency to identify effective non-pharmacological modalities for pain management across all patient populations. Distraction is a behavior management method used during procedures that may be painful or uncomfortable (2). The rationale is to reduce a patient's attention from cultivating pain signals and to thus diminish the pain experience (3).

In recent years, virtual reality (VR) has emerged as a potential analgesic and anxiolytic for medical procedures in both adult and pediatric populations (1). Virtual reality (VR) is an interactive computer-generated experience using a head-mounted display, which creates an immersive experience through visual and sound effects and enables dynamic interaction of the user in a virtual environment (2). Distraction using VR has been shown to be an effective intervention for reducing pain in children undergoing needle-related medical procedures (4). Amongst children and adolescents with kidney disease, significantly reduced pain intensity was reported during venipuncture amongst those who used VR compared to those who did not (5,6).

A randomized-control trial study conducted on pediatric orthopedics patients during out-patient procedures, Peter et al. concluded that During in-office cast and pin removal in pediatric patients, simple distraction techniques such as tablet video viewing are as effective as higher-fidelity VR headset video and interactive games in minimizing objective measures of procedural pain and subjective measures of pain and anxiety (8). On the other hand, in a study conducted on adult patients during bone marrow aspiration and biopsy procedures, Glennon et al found that More than half (51%) of the study participants reported some amount of anxiety reduction after the bone marrow aspiration and biopsy procedure, based on their reported anxiety score prior to the procedure (9). However, there is a clear lack in literature on using VR headsets in a wider patient cohort, where both adult and pediatric patients are involved.

Furthermore, in the field of otolaryngology, a randomized-control trial conducted on pediatric otolaryngology patients during nasal endoscopies, liu et al. found that VR intervention was associated with significantly reduced pain, significantly increased procedural satisfaction for patients, and significantly reduced anxiety levels for both patients and their caregivers (7). However, in addition to the study being limited to the pediatric age group, the study was also limited in terms of in-office procedures included. Therefore, further studies are warranted to apply the use of VR as an analgesic and anxiolytic to additional pediatric otolaryngology procedures in the office and peri-operative settings, as well as applying VR to additional age groups.

A randomized crossover trial was conducted on 82 adult patients who required office-based postoperative nasal endoscopy and debridement following functional endoscopic sinus surgery (FESS). Patients received either standard topical analgesia or VR treatment during nasal endoscopy and debridement, with outcomes measured using visual analog scales (VAS) for pain, Subjective Units of Distress Scale (SUDS) for anxiety, procedural time, reflexive head movements, and patient satisfaction scores. Results showed that VR treatment significantly decreased anxiety levels and reflexive head movements compared to standard treatment at the first postoperative visit. However, there were no significant differences in pain levels or procedural satisfaction between the two groups. At the second postoperative visit, patients who initially received standard treatment and later underwent VR treatment experienced reductions in pain, anxiety, reflexive head movements, and procedural time, while those who received VR treatment first showed no significant changes in pain or anxiety levels (10). Nonetheless, there are some limitations of the study, including potential bias due to lack of blinding, the relatively small sample size, and the restriction to adult patients undergoing postoperative sinonasal debridement in an outpatient setting. Thus, results regarding VR efficacy may not be generalizable to other procedures, settings, or patient populations.

In a randomized clinical trial conducted by Pandrangi et al. aimed at evaluating the efficacy of virtual reality (VR) in postoperative pain management following head and neck surgery, 30 hospitalized patients experiencing moderate to severe pain were enrolled. Patients were randomly allocated to receive either a 15-minute interactive VR gaming session using a headset or a similar gaming experience on a handheld smartphone device (control group). Pain scores were assessed before and after the intervention, alongside monitoring of opioid use. The findings revealed notable reductions in post-intervention pain among patients in the VR group immediately after the intervention and persisting for up to 3 hours afterward. Additionally, patients in the VR group displayed decreased opioid use for up to 8 hours post-intervention. Patient satisfaction with the VR intervention was high, indicating its potential as a non-pharmacologic adjunct for postoperative pain management after head and neck surgery (11).

The integration of virtual reality (VR) technology holds significant promise as a non-pharmacological method for managing pain and reducing anxiety in otolaryngology care. While existing research demonstrates overall favorable outcomes, it is often limited by small sample sizes, narrow age demographics, and specific otolaryngology interventions. Therefore, high-quality comprehensive studies involving larger sample sizes, diverse age groups and a wider array of otolaryngological interventions is warranted to establish the efficacy and feasibility of VR interventions in otolaryngology practice. This randomized controlled trial aims to contribute to this knowledge gap by investigating the impact of VR head-mounted displays on patient experiences, pain levels, and cooperation during procedures conducted at otolaryngology clinics.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged between 18-70 years old.
2. Both genders.
3. Scheduled for a nasal procedure using a 0-degree nasal endoscope.
4. Procedure performed by consultant-level rhinologists blinded to the study group assignment (VR or control group).

Exclusion Criteria:

1. History of significant nasal pathology (e.g. ciliary dyskinesia).
2. Pregnancy or breastfeeding.
3. Known neurological conditions that may affect pain perception or reported history of low pain threshold.
4. Inability to understand or follow study procedures due to language barrier or cognitive impairment.
5. Pre-existing psychiatric disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
Pain improvement | Immediately upon rhinoscopy
  VR arm will experience less pain. VR could provide a safe non-pharmacological treatment for reducing pain and improving comfort of patients, thus raising the quality of care in otolaryngology clinics, Pain scores will be measured using the Numeric Rating Pain

SECONDARY OUTCOMES:
Patient satisfaction | Immediately upon rhinoscopy
  Patient satisfaction to be measured using a 5-point Linkert scale. VR could provide a safe non-pharmacological treatment for improving comfort of patients, thus raising the quality of care in otolaryngology clinics, 1. Patient satisfaction to be measured using a 5-point Linkert scale
patient willingness to use VR in future procedures | Immediately upon rhinoscopy
  2. Patient willingness to use VR in future procedures to be measured using a 5-point Linkert scale. VR could provide a safe non-pharmacological treatment for improving comfort of patients, thus raising the quality of care in otolaryngology clinics, 2. Patient willingness to use VR in future procedures to be measured using a

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital and Research center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided